CLINICAL TRIAL: NCT01701375
Title: A Phase I and Pharmacodynamic Trial of Timed Sequential Administration of the Cyclin Dependent Kinase 4/6 Inhibitor PD 0332991 Followed by Cytarabine Plus Mitoxantrone for Adults With Relapsed and Refractory Acute Leukemias and High-Risk Myelodysplasias
Brief Title: A Phase 1 Trial of TST of PD 0332991 Followed by Cytarabine and Mitoxantrone for Adults With Relapsed and Refractory Acute Leukemias and High-Risk Myelodysplasia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Material sponsor withdrew support
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1275; NA_00076003 (Other: JHMIRB)
Record Dates: First submitted 2012-09-11; First posted 2012-10-05 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Relapsed Acute Leukemia; Refractory Acute Leukemia; High-Risk Myelodysplasia
MeSH Terms: interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): * PD 0332991 will be given orally days 1,2,3
  * Cytarabine (ara-C) will be given by continuous 72 hour intravenous infusion beginning on day 6
  * Mitoxantrone will be given over 2 hour infusion day 9, 12 hours after the completion of the ara-C infusion. The mitoxantrone dose may be reduced by 25-50% for patients who have received previous anthracyclines as determined by total previous anthracycline dose
  Interventions: Drug: PD 0332991

INTERVENTIONS:
Drug: PD 0332991 — • PD 0332991 will be given orally days 1,2,3

SUMMARY:
1.1 Primary Objectives

* To determine the feasibility, tolerability, and toxicities of administering the selective CDK 4/6 inhibitor PD 0332991 prior to the combination of ara-C and Mitoxantrone for adults with relapsed and refractory acute leukemias and high risk myelodysplasias (MDS), including primary refractory disease
* To determine the direct cytotoxic effects of single agent PD 0332991 on malignant blasts
* To determine the maximal tolerated dose (MTD) of PD 0332991 in timed sequential combination with ara-C and Mitoxantrone
* To determine if the timed sequential combination of PD 0332991 with ara-C and mitoxantrone can induce clinical responses in adults with relapsed or refractory acute leukemias and high-risk MDS

1.2 Secondary Objectives:

* To determine the ability of PD 0332991 to directly induce apoptosis in malignant cell populations in vivo
* To obtain pharmacodynamic (PD) data regarding the ability of PD 0332991 to arrest malignant cells in the G 1 phase of cell cycle, followed by synchronized release of those cells into S phase upon discontinuation of PD 0332991 and resultant enhanced ara-C cytotoxicity

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥ 18 years

  * Multilineage bone marrow failure
  * Serum creatinine ≤ 2.0 mg/dl
  * Hepatic enzymes (AST, ALT) ≤ 3x upper limit of normal (ULN)
  * Bilirubin ≤ 2.0 mg/dl, unless due to Gilbert's disease, hemolysis or leukemic infiltration
  * Left ventricular ejection fraction ≥ 45%
  * QTc ≤ 470 msec
  * RB expression is required for the action of PD 0332991. Because rb deletions and mutations are rare in acute leukemias and MDS, screening for RB expression will not be required before enrollment. Pretreatment biopsies will be stored and analyzed for RB expression if needed subsequently.

Exclusion Criteria:

* • No more than 5 cytotoxic regimens

  * Previous allogeneic or autologous stem cell transplantation permitted
  * ≥ 3 weeks delay from prior cytotoxic chemotherapy or radiation therapy
  * ≥ 2 week delay from prior biologic therapies including hematopoietic growth factors and vidaza or decitabine
  * If using Hydroxyurea, steroids, tyrosine kinase/src kinase inhibitors, arsenic, interferon for count control, must be off therapy for ≥ 48 hours prior to beginning PD 0332991
  * No concomitant use of potent CYP450 3A4 inhibitors (e.g. triazole antifungal agents) or inducers (e.g. omperazole, dilantin, dexamethasone) within 7 days prior to beginning PD 0332991

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Karp, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Weill Cornell Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 subjects were accrued
Groups:
- Arm 1: * PD 0332991 125 was given orally days 1,2,3
  * Cytarabine (ara-C) will be given by continuous 72 hour intravenous infusion beginning on day 6
  * Mitoxantrone will be given over 2 hour infusion day 9, 12 hours after the completion of the ara-C infusion. The mitoxantrone dose may be reduced by 25-50% for patients who have received previous anthracyclines as determined by total previous anthracycline dose
Period: Overall Study
Arm/Group | Arm 1
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.5 (27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Toxicities of Administration of PD 0332991 in Combination With Cytarabine and Mitoxantrone.
Description: The number of participants experiencing toxicities of administration of PD 0332991 in combination with cytarabine and mitoxantrone will be measured according to NCI-Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: 42 days
Measure: Number; unit: participants
Arm/Group | Arm 1
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: To Determine the Maximal Tolerated Dose (MTD) of PD 0332991 in Timed Sequential Combination With Ara-C and Mitoxantrone
Description: Dose escalation decisions will be based on nonhematologic toxicities in Cycle 1 (28 days) and hematologic toxicities, in the case of an aplastic marrow through Day 56, For cytopenias including ANC < 500/mm3 or platelets < 50, 000/mm3 a bone marrow will be performed between days 42 and 49.. Dose limiting toxicity (DLT) will be measured according to NCI-Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: 42 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=2)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=2)
mucositis (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes